CLINICAL TRIAL: NCT06625697
Title: Mindfulness Training and Respiration Biosignal Feedback - Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Equa Health (Industry)
Collaborators: Worcester Polytechnic Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Creswell, Co-Founder, Chief Science Officer, Equa Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11744; 1R44MH134709-01A1 (NIH)
Record Dates: First submitted 2024-09-25; First posted 2024-10-03 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Psychological Distress; Develop a Respiration Biosignal Feedback Algorithm; Utilize Respiration Algorithm to Predict Mindfulness Skills
Keywords: respiration biosignal feedback; young adults; mental health; well-being; mindfulness skills; psychological distress
MeSH Terms: conditions — Psychological Well-Being | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Respiration Biosignal Feedback Condition (Experimental): Participants will complete guided seated Equa training lessons on a laboratory smartphone device while physiological measures are tracked. After training lessons, a respiration biosignal feedback chart will appear.
  Interventions: Behavioral: Mindfulness Meditation

INTERVENTIONS:
Behavioral: Mindfulness Meditation — Participants will be instructed on how to wear the physiological monitoring equipment during the 14-unit mindfulness meditation curriculum. Participants will then complete 2-10 minute guided seated Equa training lessons on a laboratory smartphone device while physiological measures are tracked. After training lessons, a respiration biosignal feedback chart will appear on the smartphone screen. Participants will also complete a brief mindfulness survey before and after training lessons.

SUMMARY:
The goal of this research is to develop a new breathing feature on the meditation app, Equa, to help young adults who are distressed, understand their physiological responses and mindfulness skill development during meditation.

Our main aims are to build an algorithm that can use physiologic signals to:

* Give feedback about how participant physiology is changing during guided lessons on the meditation app, Equa
* Measure how much participant mindfulness skills are improving

Participants will:

* Complete a survey about demographics, their thoughts and feelings before and after the mindfulness meditation program
* Complete 14 smartphone guided mindfulness meditation training units while physiological measures are being recorded
* Complete a few brief questionnaires before and after mindfulness practices to understand potential changes in their mindfulness skills

DETAILED DESCRIPTION:
Investigators will recruit young adults to participate in a study to examine the effectiveness of respiration dynamics during meditation through phone motion data and microphones within headphones. Interested participants who contact us will be screened on study inclusion/exclusion criteria: (1) aged 18-30 years, (3]2) interested in coming on site to complete 14 smartphone guided mindfulness meditation training units, (4) willing to wear physiological monitoring equipment and provide ratings of their training experience, (5) Not currently pregnant and (6) no current or previous diagnosis of psychosis or schizophrenia

Participants are told they are going to participate in a study that focuses on monitoring physiological responses during meditation. At the start of the study, participants will complete questions via an online survey focused on demographics, prior meditation experience, their thoughts and feelings as these may be informative to participants' meditation experience.

Participants will complete a few brief questionnaires before and after each mindfulness practices to understand potential changes in mindfulness . Participant physiological data will be recorded (E.g., heart rate) via smartphones and headphones to track physiologic dynamics. Additionally, the sensory shirt, made by Hexoskin Smart Sensors; AI, will also continuously measure physiologics via two inductive plethysmography (RIP) sensors. The Hexoskin shirt also tracks motion via a three-axis accelerometer. These measures will enable investigators to better understand mindfulness measures during meditation.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-30 years of Age
* Fluent in English
* Psychological distress
* Willing to participate in guided meditation or stress management training.
* Willing and able to wear earbud headphones and a shirt which uses sensors to track motion and physiological measures.
* Willing to provide ratings on their training experience

Exclusion Criteria:

* Currently pregnant
* Current or previous diagnosis with psychosis or schizophrenia

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Optimization of deep learning algorithms that correlate changes in respiration dynamics during meditation training to changes in mindfulness skills from pre-training to post-training | Same day, change from pre-mindfulness meditation training to post-mindfulness meditation training
  Prediction accuracy of greater than 90%. There are three distinct mindfulness skills that will be measured before and after trainings - Concentration, Sensory Clarity, and Equanimity. Participants will respond to a likert scale from one to five. One is equivalent to a poor perceived level of skill and five indicates an excellent perceived level of skill.

SECONDARY OUTCOMES:
User satisfaction with the mindfulness meditation app, Equa as assessed by the Systems User Satisfaction scale at post treatment | End of treatment session at up to week 4
  Participants respond to the usability of a system by indicating the degree to which they agree or disagree with 10 statements using a 5-point scale that ranges from 1 "Strongly Disagree" to 5 "Strongly Agree" to 4 always.
User satisfaction with the mindfulness meditation app, Equa as assessed by the Mobile App Rating Scale at post treatment | At the end of treatment session at up to week 4
  The rating scale assesses app quality on four dimensions - Engagement, Functionality, Aesthetics, Information, and Subjective Quality. We are assessing Engagement and Subjective Quality only. All items are rated on a 5-point scale from "1.Inadequate" to "5.Excellent". Ratings for individual items are averaged within the applicable dimension.
Change from Baseline in total anxiety as assessed by the General Anxiety Disorder, 7-item questionnaire at post treatment | From enrollment to the end of treatment at up to week 4
  Participants respond to a questionnaire asking about how often they have been bothered by any of the listed problems over the last 2 weeks. Zero is equivalent to not at all and 3 indicates nearly every day
Change from Baseline in total depression as assessed by the Patient Health Questionnaire-9 at post treatment | From enrollment to the end of treatment at up to week 4
  Participants respond to a questionnaire asking about how often they have been bothered by any of the listed problems over the last 2 weeks. Zero is equivalent to not at all and 3 indicates nearly every day
Change from Baseline in total affect as assessed by the Positive and Negative Affect Scale at post treatment | from enrollment to the end of treatment at up to week 4
  Participants respond to a questionnaire asking to indicate the extent they have felt the following ways over the past 2 weeks. One is equivalent to not at all and five indicates extremely.
Change from Baseline in mean state mindfulness as assessed by the Mindful Attention Awareness Scale - state at post treatment | From enrollment to the end of treatment at up to week 4
  Participants respond to a questionnaire asking to what degree they were having each experience described over the past 2 weeks. Zero is equivalent to not at all and six indicates very much.
Change from Baseline in total perceived stress as assessed by the Perceived Stress Scale at post treatment | From enrollment to the end of treatment at up to week 4
  Participants respond to a questionnaire asking about their feelings and thoughts over the past 2 weeks. Zero is equivalent to never and four indicates very often.
Change from Baseline in total social well-being as assessed by the Satisfaction with Life Scale at post treatment | From enrollment to the end of treatment at up to week 4
  Participants indicate how much they agree or disagree with each of the 5 items using a 7-point scale that ranges from 7 strongly agree to 1 strongly disagree. A score of 5-9 indicates extreme dissatisfaction and a score of 31-35 indicates extreme satisfaction.
Change from Baseline in total loneliness as assessed by the UCLA Loneliness scale at post treatment | From enrollment to the end of treatment at up to week 4
  Participants indicate how often they feel the way described in each of the 20 statements using a 4-point scale that ranges from 1never to 4 always. The scoring is continuous.

CONTACTS AND LOCATIONS:
Overall Officials: David Creswell, PhD, Principal Investigator — Equa Health
Locations (1):
- GATF Building, 4615 Forbes Avenue, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will only share de-identified data from our studies that allows outside groups to independently validate our claims in our published scientific articles. All data and documentation will be de-identified and will be consistent with applicable laws and regulations.
Supporting Information: Study Protocol, ICF
Time Frame: We will provide data within six months of any approved request.
Access Criteria: Scientific groups who aim to validate our findings can make requests for data access. The study team agrees that the names and Institutions of persons either given or denied access to the data, and the bases for such decisions, will be summarized in the annual progress reports.